CLINICAL TRIAL: NCT00023946
Title: A Phase II Trial Of The Epothilone B Analog BMS-247550 (NSC 710428D) In Patients With Hepatobiliary Cancer
Brief Title: BMS-247550 in Treating Patients With Liver or Gallbladder Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02407; NCI-2012-02407 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000068878; NCI-3656; UCCRC-11045; UC#11045A (Other: University of Chicago); 3656 (Other: CTEP); P30CA014599 (NIH); N01CM62201 (NIH)
Record Dates: First submitted 2001-09-13; First posted 2003-01-27 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2012-12

CONDITIONS: Adult Primary Cholangiocellular Carcinoma; Adult Primary Hepatocellular Carcinoma; Advanced Adult Primary Liver Cancer; Cholangiocarcinoma of the Extrahepatic Bile Duct; Cholangiocarcinoma of the Gallbladder; Localized Extrahepatic Bile Duct Cancer; Localized Gallbladder Cancer; Localized Resectable Adult Primary Liver Cancer; Localized Unresectable Adult Primary Liver Cancer; Recurrent Adult Primary Liver Cancer; Recurrent Extrahepatic Bile Duct Cancer; Recurrent Gallbladder Cancer; Unresectable Extrahepatic Bile Duct Cancer; Unresectable Gallbladder Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Bile Duct Neoplasms; Gallbladder Neoplasms | interventions — ixabepilone

ARMS (1):
- Treatment (ixabepilone) (Experimental): Patients receive BMS-247550 IV over 3 hours on day 1. Treatment repeats every 21 days for at least 2 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: ixabepilone; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: ixabepilone — Given IV
  Other Names: BMS-247550; epothilone B lactam; Ixempra
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Phase II trial to study the effectiveness of BMS-247550 in treating patients who have liver or gallbladder cancer. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the objective response rate of patients with hepatobiliary cancer treated with BMS-247550.

II. Determine the toxicity of this drug in these patients. III. Determine the duration of response, median and overall survival, and time to progression in patients treated with this drug.

OUTLINE: This is a multicenter study.

Patients receive BMS-247550 IV over 3 hours on day 1. Treatment repeats every 21 days for at least 2 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed every 6 weeks until disease progression

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed locally advanced, metastatic, or recurrent hepatobiliary cancer

  * Liver (hepatocellular)
  * Bile duct (cholangiocarcinoma)
  * Gallbladder
* At least 1 unidimensionally measurable lesion

  * At least 20 mm by conventional techniques OR at least 10 mm by spiral CT scan
  * The following are not considered measurable lesions:

    * Lesions seen on colonoscopic examination or barium studies
    * Bone metastases
    * CNS lesions
    * Ascites
* No brain metastases
* Performance status - ECOG 0-2
* At least 3 months
* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Bilirubin no greater than 1.5 mg/dL
* AST/ALT no greater than 2.5 times upper limit of normal
* Creatinine no greater than 1.5 mg/dL
* Creatinine clearance at least 60 mL/min
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* No grade 2 or greater peripheral neuropathy
* No other uncontrolled concurrent illness
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study compliance
* No prior allergic hypersensitivity reaction attributed to compounds containing Cremophor EL (e.g., paclitaxel or compounds of similar chemical or biological composition to BMS-247550)
* No other currently active malignancy except nonmelanoma skin cancer, carcinoma in situ of the cervix, or cancer for which patient has completed therapy and is at less than 30% risk of relapse
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No concurrent immunotherapy
* No prior chemotherapy
* No other concurrent chemotherapy
* No concurrent hormonal therapy
* No concurrent therapeutic radiotherapy
* At least 30 days since prior investigational agents
* At least 7 days since prior cimetidine
* No concurrent cimetidine
* No other concurrent commercial or investigational anticancer agents or therapies
* No concurrent unconventional therapies, food, or vitamin supplements (e.g., St. John's Wort)
* No concurrent combination antiretroviral therapy for HIV-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2001-08; Primary Completion 2005-07 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Objective response rate (partial or complete response) evaluated by RECIST | Up to 8 years
  A 10% response rate precludes further study whereas a 25% response rate would indicate that further study is warranted.
Frequency and extent of cytotoxic activity graded according to the NCI CTC Version 2.0 | Up to 8 years
Time to disease progression | From the first day of treatment until the date PD or death is first reported, assessed up to 8 years
  Will also be evaluated using the Kaplan-Meier estimator.
Overall survival | From the time measurement criteria are met for CR/PR (whichever is first recorded) until the first date that PD is objectively documented, assessed up to 10 years
  Will also be evaluated using the Kaplan-Meier estimator.

CONTACTS AND LOCATIONS:
Overall Officials: Hedy Kindler, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States